CLINICAL TRIAL: NCT01952795
Title: Effect of Hypocaloric Diet and Exercise in Obese Women Who Are Subjected to IVF Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-DHE-2011-42
Record Dates: First submitted 2013-09-23; First posted 2013-09-30 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diet and exercise (Active Comparator): Total caloric intake aimed at maintaining a diet with> 50% of the caloric content in the form of carbohydrates, less than 10% in the form of saturated fats and 20% from monounsaturated / polyunsaturated (if applicable, up to 25% fat monounsaturated), less than 300 mg / day of dietary cholesterol and about 1.0 g of protein / kg ideal body weight / day. 3 sessions per week on a bicycle ergometer or on a treadmill (according to body fat distribution and other parameters) modifications carried out weekly, with a gradual increase as to exercise until maximal oxygen consumption 60 - 70% would always preceded by heating 5 minutes.
  Interventions: Behavioral: Diet and exercise
- No intervention (No Intervention): Usual diet and exercise

INTERVENTIONS:
Behavioral: Diet and exercise — Total caloric intake aimed at maintaining a diet with> 50% of the caloric content in the form of carbohydrates, less than 10% in the form of saturated fats and 20% from monounsaturated / polyunsaturated (if applicable, up to 25% fat monounsaturated), less than 300 mg / day of dietary cholesterol and about 1.0 g of protein / kg ideal body weight / day.
  Arms: Diet and exercise

SUMMARY:
The purpose of this study is to determine the impact of diet and physical exercise program on pregnancy rate and live birth in obese women who undergo an IVF cycle.

DETAILED DESCRIPTION:
The objective of this study is showing that obesity significantly affects the in vitro fertilization cycles lowering the reproductive capacity. The study is been performed in Hospital de la Santa Creu i Sant Pau and Fundació Puigvert of Barcelona. Patients recluted are obese women with sterility problems that require in vitro fertilization (IVF) with a body mass index BMI between 30-35. It´s a randomised study in which half of the patients undergo to a 6 weeks program of diet and exercice. We will analyse the response to ovaric stimulation, the results of the egg retrieval (ovocyte number and quality), rates of fecundation, embryo implantation and clinical gestation.

ELIGIBILITY:
Inclusion Criteria:

* Women who want pregnancy.
* Basal FSH levels ≤ 10 IU / l.
* Infertility to justify treatment with IVF/ICSI.
* Being included in a long protocol with GnRH agonist.
* Presence of both ovaries and uterus able to support embryo implantation and pregnancy.
* Body mass index (BMI) ≥ 30 kg/m2 and ≤ 35 kg/m2.
* Absence of pregnancy before starting ovarian stimulation.
* Having given their written consent.

Exclusion Criteria:

* Female age ≤ 18 years and ≥ 35 years.
* Severe male factor not permit an IVF-ICSI with ejaculated sample.
* Patients with low ovarian reserve (basal FSH levels ≥ 10 IU / l or lower antral follicle count to 6 follicles in both ovaries).
* HIV seropositivity, HBV or HCV.
* Clinically important disease.
* Having frozen embryos from previous cycles of assisted reproduction.
* Unexplained vaginal bleeding.
* Poor response in previous IVF cycles with standard stimulation protocols
* Any contraindication to become pregnant.
* Known allergy to preparations of gonadotropins or its excipients.
* High consumption of alcohol, drugs or psychotropic drugs.
* Concurrent participation in another study.
* Patients who have done previous cycles of IVF / ICSI without success

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 14 days after embryo transfer
  Pregnancy rate by cycle

SECONDARY OUTCOMES:
Hyperstimulation rate | At luteal phase and first weeks of pregnancy
  Number of patients with moderate or severe hyperstimulation
Fertility rate | 24 hours post pick up
  Rate of mature oocytes fertilized by conventional IVF or ICSI
Mature oocytes | Pick up day
  Number of total mature oocytes obtained after stimulation
Cancellation rate | Durinf the stimulation in follicular phase
  Stimulated Patients who fail to perform the follicular puncture
Good quality embryos | Day 3 to 5 post pick up
  Number of good quality embryos obtained (A and B) by patient
Abortion rate | First trimester of pregnancy
  Number of non evolutive pregnancies during the first trimester
Live birth rate | Between 7 a 9 months after treatment
  Amount of patients who finish the treatment with a live newborn

OTHER OUTCOMES:
Leptin, adiponectin, resistin, interleukin VI, TNF-α, visfatin, IGF1 and PAI I | During the stimulation phase
  Study the relationship between obesity and measurable surrogate parameters the same as the products of secretion of fat (leptin, adiponectin, resistin, interleukin VI, TNF-α, visfatin, IGF1 and PAI I) or with inflammatory parameters results of an IVF cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Espinós-Gómez, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain